CLINICAL TRIAL: NCT03891914
Title: Prospective Comparison of 18F-choline PET/CT and 18F-FDG PET/CT in the Initial Work-up of Multiple Myeloma
Acronym: MYELOCHOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/32
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Myeloma Multiple
Keywords: Multiple Myeloma; PET/CT; 18F-FDG; 18F-FCH
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptomatic Multiple Myeloma on first-line treatment (Experimental)
  Interventions: Drug: Positron Emission Tomography using 18F-FCH; Drug: Positron Emission Tomography using 18F-FDG

INTERVENTIONS:
Drug: Positron Emission Tomography using 18F-FCH — Positron Emission Tomography imaging coupled with scanner (PET-CT). with the injection of a radiopharmaceutical drug, the 18F-FCH(or fluorocholine) for the detection of bone lesions
Drug: Positron Emission Tomography using 18F-FDG — Positron Emission Tomography imaging coupled with scanner (PET-CT). with the injection of a radiopharmaceutical drug, the 18F-FDG (or fluorodeoxyglucose) for the detection of bone lesions

SUMMARY:
Multiple myeloma (MM) survival has been improved during the last decade owing to new treatments. Hence, it has become a matter of importance to precisely define the depth of MM response to therapy. 18F-FDG PET/CT (FDG-PET) has proved to be superior to X-rays for the initial staging of MM. It is now recommended by the International Myeloma Working Group (IMWG) during the initial work-up and for response evaluation, as it is superior to MRI in that setting. However, sensitivity of FDG-PET remains inferior to that of MRI for the initial staging of MM. Indeed, FDG-PET remains limited for the evaluation of skull lesions (due to brain physiological background) or spine infiltrative disease. Therefore, there is a need for a new diagnostic tool which could have equivalent sensitivity to that of MRI at diagnosis, and could bring better baseline information than FDG PET for therapy evaluation. Ultimately, this tool would be a one-stop-shop exam for diagnosis and patient follow-up during treatment. 18F-Choline, a tracer of phospholipids of cell membrane, has shown potential as compared to 18F-FDG in a recent retrospective study, with about 70% more lesions detected in MM patients with suspected relapsing disease. Following that perspective, our main objective is to compare prospectively, in a cohort of newly diagnosed MM, the detection rate of MM lesions by 18F-Choline PET/CT (FCH-PET) vs. FDG-PET. Our secondary objectives will be to compare the performance of both PET modalities as regard to MRI as well as the detection rate of extra-medullary lesions. Patients with MM will proceed to FCH-PET, FDG-PET and then Whole-Body MRI within 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Multiple Myeloma on first-line treatment as defined by 2014 International Myeloma Working Group criteria
* Measurable disease either by serum or urinary monoclonal protein level or by serum free light chains assay
* Age > 18 years old at time of signed consent
* Beneficiary of social security insurance
* Signed informed consent

Exclusion Criteria:

* Previous Multiple Myeloma treatment
* Previous cancer with less than 5 year of complete remission (including plasmacytoma)
* Chemotherapy in the 6 months preceding the inclusion
* Uncontrolled diabetes mellitus
* Medullary growth factor injection less than 48 hours before imaging procedures
* Ongoing corticosteroid therapy, or given less than 72 hours before PET-CT imaging
* Pregnant or nursing (lactating) women
* Childbearing potential woman without adequate barrier contraception method (HAS criteria)
* Freedom deprivated patient by judiciary or administrative decision
* Patient under legal protection or unable to express its own consent
* PET contraindication (known allergy to 18F-FCH or 18F-FDG or excipient)
* MRI contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of whole-body bone lesions | Day 0
  The numbers of bone lesions detected by 18F-FCH PET-CT and that are suspected to be related to multiple myeloma, will be counted. Every bone lesion will be validated by the reference test which is composed of MRI standard sequences plus whole-body diffusion MRI. A bone lesion that is not present on MRI but is present on any of the PET modalities must be validated by an expert multidisciplinary consensus.
Number of whole-body bone lesions | Day 7
  The numbers of bone lesions detected by 18F-FDG PET-CT, and that are suspected to be related to multiple myeloma, will be counted. Every bone lesion will be validated by the reference test which is composed of MRI standard sequences plus whole-body diffusion MRI. A bone lesion that is not present on MRI but is present on any of the PET modalities must be validated by an expert multidisciplinary consensus.
Number of bone lesions within defined skeletal areas | Day 0
  Six skeletal areas are defined : skull - spine - pelvis - sternum and ribs - superior limbs - inferior limbs. The number of bone lesions that are suspected to be related to myeloma in each of these skeletal area is assessed on 18F-FCH PET-CT Every bone lesion will be validated by the reference test which is composed of MRI standard sequences plus whole-body diffusion MRI. A bone lesion that is not present on MRI but is present on any of the PET modalities must be validated by an expert multidisciplinary consensus
Number of bone lesions within defined skeletal areas | Day 7
  Six skeletal areas are defined : skull - spine - pelvis - sternum and ribs - superior limbs - inferior limbs. The number of bone lesions that are suspected to be related to myeloma in each of these skeletal area is assessed on 18F-FDG PET-CT. Every bone lesion will be validated by the reference test which is composed of MRI standard sequences plus whole-body diffusion MRI. A bone lesion that is not present on MRI but is present on any of the PET modalities must be validated by an expert multidisciplinary consensus

SECONDARY OUTCOMES:
Diagnostic performance for the detection of focal bone lesions | Day 0
  Sensitivity, specificity, positive predictive value, negative predictive value and accuracy of 18F-FCH PET-CT will be calculated based on two different reference test. First reference test will be standard MRI sequences (T1SE, T2-STIR). Second reference test will be composed of standard MRI sequences plus whole-body diffusion MRI acquisitions.
Diagnostic performance for the detection of focal bone lesions | Day 7
  Sensitivity, specificity, positive predictive value, negative predictive value and accuracy of 18F-FDG PET-CT will be calculated based on two different reference test. First reference test will be standard MRI sequences (T1SE, T2-STIR). Second reference test will be composed of standard MRI sequences plus whole-body diffusion MRI acquisitions.
Diagnostic performances for the detection of diffuse infiltrative disease of the spine | Day 7
  Sensitivity, specificity, positive predictive value, negative predictive value and accuracy of 18F-FDG PET-CT will be calculated based on standard MRI sagittal acquisitions of the spine.
Diagnostic performances for the detection of diffuse infiltrative disease of the spine | Day 0
  Sensitivity, specificity, positive predictive value, negative predictive value and accuracy of 18F-FCH PET-CT will be calculated based on standard MRI sagittal acquisitions of the spine.
Number of extra-medullary lesions | Day 7
  Each extra-medullary lesion detected on 18F-FDG PET-CT will be validated by an expert multidisciplinary consensus
Number of extra-medullary lesions | Day 0
  Each extra-medullary lesion detected on 18F-FCH PET-CT will be validated by an expert multidisciplinary consensus

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital - Haut-Lévêque, Pessac, France

REFERENCES:
- [Derived] Mesguich C, Hulin C, Latrabe V, Asselineau J, Bordenave L, Perez P, Hindie E, Marit G. Prospective Comparison of 18F-Choline Positron Emission Tomography/Computed Tomography (PET/CT) and 18F-Fluorodeoxyglucose (FDG) PET/CT in the Initial Workup of Multiple Myeloma: Study Protocol of a Prospective Imaging Trial. JMIR Res Protoc. 2020 Sep 10;9(9):e17850. doi: 10.2196/17850. PMID 32909953